CLINICAL TRIAL: NCT05879822
Title: A Phase 2 Study Evaluating INCB099280 in Participants With Select Solid Tumors Who Are Immune Checkpoint Inhibitor Naive
Brief Title: A Study to Evaluate INCB099280 in Participants With Select Solid Tumors Who Are Immune Checkpoint Inhibitor Naive
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 99280-211; 2022-502716-37-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2023-05-19; First posted 2023-05-30 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumor
Keywords: Advanced Solid Tumor; Hepatocellular Carcinoma; Cutaneous Melanoma; PD-L1-positive NSCLC; Non-small Cell Lung Cancer; Renal Cell Carcinoma; Urothelial Cancer; MSI-H/dMMR Tumors
MeSH Terms: conditions — Carcinoma, Hepatocellular; Melanoma; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell

STUDY DESIGN:
Intervention Model Description: The study consists of 2 parts. In Part 1, participants with 6 different tumor types will be randomized 1:1:1 to INCB099280 Dose 1, INCB099280 Dose 2, or INCB099280 Dose 3 twice daily (BID). At the end of Part 1, an integrated analysis will be performed to select a dose. Once a dose is selected, Part 2 will proceed to complete enrollment for each of the 6 disease-specific cohorts at the selected dose.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: INCB099280 Dose 1 (Experimental): Participants will receive INCB099280 dose 1 twice daily (BID) for up to 2 years.
  Interventions: Drug: INCB099280
- Part 1: INCB099280 Dose 2 (Experimental): Participants will receive INCB099280 dose 2 twice daily (BID) for up to 2 years.
  Interventions: Drug: INCB099280
- Part 1: INCB099280 Dose 3 (Experimental): Participants will receive INCB099280 dose 3 twice daily (BID) for up to 2 years
  Interventions: Drug: INCB099280
- Part 2: INCB099280 Dose selected from Part 1 (Experimental): Participants will receive INCB099280 dose selected from Part 1 twice daily (BID) for up to 2 years.
  Interventions: Drug: INCB099280

INTERVENTIONS:
Drug: INCB099280 — Administered as specified in the treatment arm description

SUMMARY:
This study is being conducted to determine the safety, tolerability, and preliminary efficacy of INCB099280 in participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Immunotherapy naive and without access to approved and/or available immune checkpoint inhibitor (ICI) therapy.
* Measurable disease per RECIST v1.1.
* One of the following disease settings:

  * Unresectable or metastatic Child-Pugh Class A hepatocellular carcinoma (HCC) not eligible for surgical and/or locoregional therapy and have not received prior systemic therapy or had disease progression following primary therapy.
  * Unresectable or metastatic cutaneous melanoma and have not received more than 1 previous systemic therapy for advanced disease.
  * Unresectable Stage III PD-L1-positive (TPS ≥ 50% using the Dako PD-L1 IHC 22C3 assay) non-small cell lung cancer (NSCLC) without actionable molecular biomarkers and have not received prior systemic therapy and where chemoradiation is contraindicated; in addition, able to provide fresh or archival tumor tissue for central confirmation of PD-L1 expression.
  * Stage IV PD-L1-positive (TPS ≥ 50% using the Dako PD-L1 IHC 22C3 assay) NSCLC without actionable molecular biomarkers and have not received prior systemic therapy; in addition, able to provide fresh or archival tumor tissue for central confirmation of PD-L1 expression.
  * Relapsed or Stage IV clear cell renal cell carcinoma (RCC) after having received 1 prior systemic therapy for relapsed or Stage IV disease.
  * Cisplatin-ineligible, locally advanced or Stage IV urothelial cancer (UC) and have not received prior systemic therapy for locally advanced or Stage IV UC and able to provide fresh or archival tumor tissue for central confirmation of PD-L1 expression using the Dako PD-L1 IHC 22C3 assay.
  * Advanced or metastatic microsatellite instability high (MSI-H) or deficient mismatch repair (dMMR) (as determined by an approved assay) solid tumors and able to provide fresh or archival tumor tissue for central confirmation of MSI-H or dMMR.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Life expectancy > 3 months.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Known history of an additional malignancy.
* Central nervous system (CNS) metastases requiring treatment and/or leptomeningeal disease.
* Toxicity from prior therapy that has not recovered.
* Prior receipt of an PD-1, anti-PD-L1, or anti-PD-L2 agent or treatment with an immune modulator (eg, CTLA-4, GITR, LAG3, TIM3, OX40, ICOS, IL-2, 4-1BB, CAR-T cell).
* Received thoracic radiation within 6 months of the first dose of study treatment.
* Participation in another interventional clinical study while receiving INCB099280.
* Impaired cardiac function or clinically significant cardiac disease.
* History or evidence of interstitial lung disease including noninfectious pneumonitis.
* Presence of gastrointestinal conditions that may affect drug absorption.
* Any autoimmune disease requiring systemic treatment in the past 5 years.
* Diagnosis of immunodeficiency or receiving chronic systemic steroid therapy at a daily dose exceeding 10 mg of prednisone or equivalent.
* Active infection requiring systemic therapy.
* History of organ transplantation, including allogeneic stem cell transplantation.
* Receipt of systemic antibiotics within 28 days of first dose of study treatment.
* Probiotic usage is prohibited during screening and throughout the study treatment period.
* Received a live vaccine within 28 days of the planned start of study drug.
* Laboratory values outside the Protocol-defined ranges.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2026-07-22 (Estimated); Study Completion 2026-07-22 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  Defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR), as determined by investigator radiographic disease assessment according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to 2 years 3 months
  Defined as any Adverse event either reported for the first time or worsening of a pre-existing event after first dose of study drug up to 90 days after the last dose of study drug or until the start of new anticancer therapy, whichever occurs first.
Number of participants with TEAEs leading to dose modification or discontinuation | Up to 2 years
  Number of participants with TEAEs leading to dose modification or discontinuation.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Up to 2 years
  Defined as the percentage of participants with the best overall response of CR or PR, or stable disease (SD), after a minimum of 15 weeks following the initiation of study treatment by investigator assessment per RECIST v1.1.
Duration Of Response (DOR) | Up to 2 years
  Defined as the time from the earliest date of CR or PR until the earliest date of disease progression, as determined by investigator radiographic disease assessment according to RECIST v1.1, or death due to any cause if occurring sooner than progression.
INCB099280 pharmacokinetic (PK) in Plasma | Pre dose and 1, 2 and 6 hours post dose on Cycle 1 Day 1 and Cycle 2 Day 1. Pre dose every other cycle until Cycle 11 Day 1 (Cycle 3 Day 1, Cycle 5 Day 1, Cycle 7 Day 1, Cycle 9 Day 1 and Cycle 11 Day 1) (each cycle is 28 days)
  INCB099280 concentration in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (54):
- Brazil (13):
  - Fundacao Pio Xii Hospital de Cancer de Barretos, Barretos
  - Cionc-Centro Integrado de Oncologia de Curitiba, Curitiba
  - Hospital Erasto Gaertner - Liga Paranaense de Combate Ao Câncer, Curitiba
  - Oncosite - Centro de Pesquisa Clinica E Oncologia, Ijuí
  - Clinica de Neoplasias Litoral Ltda, Itajaí
  - Fundacao Doutor Amaral Carvalho, Jaú
  - Hospital de Cancer de Londrina, Londrina
  - Irmandade Da Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Hgb - Hospital Giovanni Battista - Mae de Deus Center, Porto Alegre
  - Hospital Ernesto Dornelles, Porto Alegre
  - Hospital Nossa Senhora Da Conceicao, Porto Alegre
  - Cepho - Centro de Estudos E Pesquisas de Hematologia E Oncologia, Santo André
  - A. C. Camargo Cancer Center, São Paulo
- The People'S Hospital of Guangxi Zhuang Autonomous Region, Nanning, China
- Georgia (12):
  - High Technology Hospital Medcenter, Batumi
  - Jsc Evex Hospitals, Kutaisi
  - Caucasus Medical Centre Llc, Tbilisi
  - Archangel St. Michael Multi Profile Clinical Hospital, Tbilisi
  - Israel-Georgian Medical Research Clinic Helsicore, Tbilisi
  - Todua Clinic, Llc, Tbilisi
  - New Hospitals, Tbilisi
  - Tim-Tbilisi Institute of Medicine Ltd, Tbilisi
  - Tbilisi State Medical University and Ingorokva High Medical Technology University Clinic, Llc, Tbilisi
  - Institute of Clinical Oncology Ltd, Tbilisi
  - Cancer Research Center Ltd, Tbilisi
  - Medulla Chemotherapy and Immunotherapy Clinic, Tbilisi
- Greece (3):
  - 251 Air Force General Hospital, Athens
  - University Hospital of West Attica - Attikon, Athens
  - Euromedica General Clinic of Thessaloniki, Thessaloniki
- Hungary (2):
  - Semmelweis Egyetem, Budapest
  - Orszagos Onkologiai Intezet, Budapest
- New Zealand (2):
  - Dunedin Hospital, Dunedin
  - Rotorua Hospital, Rotorua
- Romania (11):
  - Centrul Medical Medicover Victoria, Bucharest
  - Institutul Clinic Fundeni Clinica, Bucharest
  - Institutul Oncologic Prof. Dr. Ion Chiricuta Cluj-Napoca, Cluj-Napoca
  - Spitalul Clinic Militar de Urgenta Dr. Constantin Papilian Cluj-Napoca, Cluj-Napoca
  - Medisprof, Cluj-Napoca
  - Centrul de Oncologie Sf. Nectarie Craiova, Craiova
  - Sc Radiotherapy Center Cluj Srl, Floreşti
  - Institutul Regional de Oncologie Iasi, Iași
  - S.C. Medical Center Gral Srl, Ploieşti
  - S C Oncocenter Oncologie Medicala S R L, Timișoara
  - Oncomed Srl, Timișoara
- South Africa (5):
  - Cape Town Oncology Trials (Pty) Ltd, Cape Town
  - Johese Clinical Research: Midstream, Centurion
  - Wits Clinical Research, Johannesburg
  - The Medical Oncology Centre of Rosebank, Johannesburg
  - Phoenix Pharma (Pty) Ltd, Port Elizabeth
- Turkey (Türkiye) (5):
  - Medical Park Seyhan Hospital, Adana
  - Hacettepe University Medical Faculty, Ankara
  - Trakya University Medical Faculty, Edirne
  - Goztepe Prof. Dr. Suleyman Yalcin City Hospital, Istanbul
  - Kocaeli Universitesi Tip Fakultesi, Kocaeli

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: A Study to Evaluate INCB099280 in Participants With Select Solid Tumors Who Are Immune Checkpoint Inhibitor Naive — https://incyteclinicaltrials.com/studies/incb-99280-211